CLINICAL TRIAL: NCT01488279
Title: Effect of Sitagliptin on Short-Term Metabolic Dysregulation of Oral Glucocorticoid Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Annis Marney, MD, MSCI, Assistant Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MISP 39681
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Pre-diabetes; Impaired Fasting Glucose; Impaired Glucose Tolerance
Keywords: Pre-diabetes; Impaired fasting glucose; Impaired glucose tolerance; Steroid-induced hyperglycemia
MeSH Terms: conditions — Glucose Intolerance | interventions — Dexamethasone; Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled crossover study
Who Masked: Participant, Investigator
Masking Description: Drugs were dispensed by the pharmacy with both the patient and investigator blinded
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone 2.5mg and Sitagliptin100mg (Active Comparator): Participants received Dexamethasone 2.5 mg plus Sitagliptin 100 mg daily for 8 days
  Interventions: Drug: Dexamethasone 2.5 mg and Sitagliptin 100 mg; Drug: Dexamethasone 2.5 mg and placebo tablet
- Dexamethasone 2.5mg and placebo tablet (Placebo Comparator): Participants received Dexamethasone 2.5 mg plus Sitagliptin-matched placebo tablet daily for 8 days.
  Interventions: Drug: Dexamethasone 2.5 mg and Sitagliptin 100 mg; Drug: Dexamethasone 2.5 mg and placebo tablet

INTERVENTIONS:
Drug: Dexamethasone 2.5 mg and Sitagliptin 100 mg — Participants received Dexamethasone 2.5mg plus Sitaliptin 100mg daily for 8 days
  Other Names: Sitagliptin
Drug: Dexamethasone 2.5 mg and placebo tablet — Participants rececived Dexamethasone 2.5 mg plus placebo tablet daily for 8 days
  Other Names: Placebo

SUMMARY:
The investigators hypothesize that sitagliptin will significantly reduce impairments in insulin secretion and insulin resistance resulting from short-term oral glucocorticoid therapy.

DETAILED DESCRIPTION:
The investigators plan to conduct a prospective, randomized, double-blind, placebo-controlled parallel arm crossover study comparing insulin secretion and insulin resistance in subjects with impaired fasting glucose on oral glucocorticoid therapy + placebo versus subjects on oral glucocorticoid therapy + sitagliptin. For the oral glucocorticoid therapy, we plan to use dexamethasone (dex) 2.5 mg daily. We chose dex for known glycemic effects, improved compliance, and once daily dosing.

Previous studies have shown that in humans, glucocorticoid-induced insulin resistance develops within 4 hours with infused drug at high dose (methylprednisolone 500 mg x single infusion) and does not change with duration of drug therapy of up to 3 months.10 Furthermore, more modest doses over a short duration (dex 2.0 mg orally daily x 2 days) have been shown to decrease insulin-mediated glucose disposal.11 12 Thus, studying acute effects of oral dex at 2.5 mg daily x 7 days should be more than adequate to achieve impaired glucose-mediated insulin secretion and impaired insulin-mediated glucose disposal.

In order for sitagliptin to have the desired effect, drug should be administered for at least 7 days (5 half-lives plus 40% more for margin of error). We plan to study subjects with impaired fasting glucose or impaired glucose tolerance as they would likely be candidates for DPP-IV therapy in the future and would be likely to have impaired insulin secretion and impaired glucose disposal amenable to DPP-IV therapy.

A total of 10 participants were enrolled in this study. Participants were given 2.5 mg dexamethasone daily plus either placebo tablet or sitagliptin daily for 8 days with a washout period prior to crossover. The order of study drug administration was randomized. Participants underwent blood sampling, mixed meal testing (MMT), and intravenous glucose tolerance testing (IVGTT) before and after each study period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* impaired fasting glucose
* We will stratify for weight and age.

Exclusion Criteria:

* Known Type 2 DM
* Severe disease preventing participation in study
* On chronic steroids for any reason
* Already taking DPP-4 inhibitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annis M Marney, MD, MSCI, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont Clinical Research Center, South Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin, Then Placebo: Dex 2.5 mg + sitagliptin 100 mg daily (7 days), washout (4-6 weeks), dex + placebo (7 days)
- Placebo, Then Sitaglipton: Dex 2.5 mg + placebo (7 days), washout (4-6 weeks), Sitalgiptin + placebo ( 7 days)
Period: Overall Study
Arm/Group | Sitagliptin, Then Placebo | Placebo, Then Sitaglipton
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin, Then Placebo: This arm involves randomization to dexamethasone 2.5 mg + sitagliptin 100 mg daily x 7 days followed by MTT and IVGTT on subsequent days. There was a 4-6 week washout, then subjects crossed over to dex + placebo.
- Placebo, Then Sitagliptin: This arm involves randomization to dexamethasone 2.5 mg orally + placebo x 7 days followed by MTT and IVGTT on subsequent days. There was a 4-6 weeks washout, then subjects crossed over to dex + sitagliptin.
- Total: Total of all reporting groups
Arm/Group | Sitagliptin, Then Placebo | Placebo, Then Sitagliptin | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (5.5) | 52.5 (5.5) | 52.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin Sensitivity measured at the end of each treatment period. The primary outcome variable was the difference in the disposition index (DI) determined as the product of the acute insulin response to glucose (AIRg) x the insulin sensitivity index (SI) in subjects during IVGTT on the 8th day (after 7 days) of on dex + placebo, then a after a washout of approximately 4 weeks, participants crossed over to dex + sitagliptin 100 mg x 7 days. Subjects were randomized to order of medication. The primary analyses will be an ANCOVA, including baseline responses as a covariate.
Time Frame: Measured on day #8 (after 8 days of sitagliptin or placebo) followed by a 4 week washout then measured again on day #8 (after 8 days of crossover treatment).
Population: Subjects were randomized to the order to study medication (dex + sitagliptin vs dex + placebo) by the pharmacy in order to keep double blinding
Measure: Mean (Standard Error); unit: ratio without units
Groups:
- Sitagliptin: This arm involves randomization to dexamethasone 2.5 mg + sitagliptin 100 mg daily x 7 days followed by MTT and IVGTT on subsequent days.
- Placebo: This arm involves randomization to dexamethasone 2.5 mg orally + placebo x 7 days followed by MTT and IVGTT on subsequent days.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 10 | 10
ratio without units | 1835.4 (340.0) | 1846.0 (340.0)
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; 2X2 crossover design with baseline values. To compare the means between Sitagliptin and Placebo, a sequential three step testing process used. The results of the third step, the direct treatment comparisons are presented; Test type: Superiority; p = .983, ANOVA; Mean Difference (Net) = -10.8, 95% CI 2-sided [-1147.6 to 1126.0], Standard Error of Mean 480.8

2. Secondary Outcome: Change in Active GIP
Description: We had planned to measure the difference or change in active GIP in response to the MTT between the 2 study drug periods: on sitagliptin versus on placebo. However, when other measures were negative, we opted not to pursue this lab assay for cost and time. We did not perform measures of GIP.
Time Frame: Active GIP would have been measured during MTT after 1 week of dex + sitagliptin and again after 1 week of dex + placebo, but we did not measure active GIP
Population: We did not measure GIP
Groups:
- Placebo: This arm involves randomization to dexamethasone 2.5 mg + placebo daily x 7 days followed by MTT and IVGTT on subsequent days.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Active GLP-1
Description: As with GIP, we had planned to measure the difference or change in active GLP-1 in response to the MTT between the 2 study drug periods: on sitagliptin versus on placebo. We had hypothesized that GIP and GLP-1 would be elevated while on the DPP4 inhibitor compared to placebo as this is the mechanism of action of the drug sitagliptin. When other measures were negative, we elected not to pursue this due to time and cost.
Time Frame: Active GLP-1 would have been measured during MTT after 1 week of dex + sitagliptin and again after 1 week of dex + placebo, but we did not measure active GLP-1
Population: We did not measure GLP-1
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Glucose Response
Description: Change in glucose response during the MTT. This was the Si (insulin sensitivity). We sought to determine whether there was an improvement in the glucose response after a meal on the DPP4i compared to placebo in the face of steroid (dexamethasone).
Time Frame: measured on day #9 (after 7 days of study drug and 1 day of IVGTT) of sitagliptin during MTT, then after 4 week washout, measured again on day #9 (after 7 days of study drug + 1 day of IVGTT) of dex + placebo during MTT
Measure: Least Squares Mean (Standard Error); unit: response x 10000 / minute / microUnit/ml
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 10 | 10
response x 10000 / minute / microUnit/ml | 4.219 (1.368) | 4.228 (1.368)
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority; p = .997, ANOVA; Mean Difference (Net) = -0.008, 95% CI 2-sided [-4.585 to 4.568], Standard Error of Mean 1.935

5. Secondary Outcome: Change in Insulin Secretion (AIRg or Acute Insulinogenic Response to Glucose)
Description: We measured the change in insulin secretion (AIRg or acute insulinogenic response to glucose) during the MTT and compared the insulin secretion on the DPP4 inhibitor (sitagliptin) compared to placebo. We had expected the AIRg to be greater with DPP4i compared to placebo.
Time Frame: measured twice: on day #8 (after 7 days of study drug and 1 day of IVGTT) of sitagliptin during MTT, then after 4 week washout, measured again on day #8 (after 7 days of study drug + 1 day of IVGTT) of dex + placebo during MTT
Measure: Least Squares Mean (Standard Error); unit: pmol/l
Groups:
- Sitagliptin: Participants received dex 2.5 mg + sitagliptin 100 mg daily x 7 days.
- Placebo: Participants received dex 2.5 mg + placebo daily x 7 days.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 10 | 10
pmol/l | 519.6 (0.460) | 558.6 (35.3)
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority; p = .460, ANOVA; Mean Difference (Net) = -38.9, 95% CI 2-sided [-156.9 to 79.0], Standard Error of Mean 49.9

ADVERSE EVENTS:
Time Frame: Only during the study period (approximately 6-10 weeks per subject). Each participant had 2 weeks of study drug total plus around 4 weeks of washout.
Groups:
- Sitagliptin, Then Placebo: This arm involves randomization to dexamethasone 2.5 mg + sitagliptin 100 mg daily x 7 days followed by MTT and IVGTT on subsequent days.
  Dexamethasone medication: 2.5 mg daily dexamethasone x 7 days
- Placebo, Then Sitagliptin: This arm involves randomization to dexamethasone 2.5 mg orally + placebo x 7 days followed by MTT and IVGTT on subsequent days
  Dexamethasone medication: 2.5 mg daily dexamethasone x 7 days
Arm/Group | Sitagliptin, Then Placebo | Placebo, Then Sitagliptin
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Sample size or length of study drug may have been too small

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less